CLINICAL TRIAL: NCT04780308
Title: How Many K Wires do we Need in the Surgical Treatment of Pediatric Type III Supracondylar Humeral Fracture?
Brief Title: Pediatric Type III Supracondylar Humeral Fracture
Acronym: Fracture
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Alkan Bayrak, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 2014/18/05
Record Dates: First submitted 2021-02-07; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Supracondylar Humerus Fracture; Pediatric Fractures
Keywords: pediatric; supracondylar humeral fracture; k wires; closed reduction; pin configuration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1 medial 1 lateral K-wire: Pediatric Gartland Type 3 supracondylar humeral fractures fixed by 1 medial 1 lateral K-wire
  Interventions: Procedure: Pediatric Garthland Type 3 supracondylar humeral fractures fixed by K-wires
- 1 medial 2 lateral K-wire: Pediatric Gartland Type 3 supracondylar humeral fractures fixed by 1 medial 2 lateral K-wire
  Interventions: Procedure: Pediatric Garthland Type 3 supracondylar humeral fractures fixed by K-wires
- 2 medial 1 lateral K-wire: Pediatric Gartland Type 3 supracondylar humeral fractures fixed by 2 medial 1 lateral K-wire
  Interventions: Procedure: Pediatric Garthland Type 3 supracondylar humeral fractures fixed by K-wires
- 2 lateral K-wire: Pediatric Gartland Type 3 supracondylar humeral fractures fixed by 2 lateral K-wire
  Interventions: Procedure: Pediatric Garthland Type 3 supracondylar humeral fractures fixed by K-wires
- 3 lateral K-wire: Pediatric Gartland Type 3 supracondylar humeral fractures fixed by 3 lateral K-wire
  Interventions: Procedure: Pediatric Garthland Type 3 supracondylar humeral fractures fixed by K-wires

INTERVENTIONS:
Procedure: Pediatric Garthland Type 3 supracondylar humeral fractures fixed by K-wires — The effects of the different types of K-wire configuration on Pediatric Gartland Type 3 supracondylar humeral fractures were evaluated. Pediatric Gartland Type 3 supracondylar humeral fractures operated under general anesthesia with open or closed reduction. After reduction checked by fluoroscopy K-wires applied in different configurations.

SUMMARY:
The purpose of this study was to compare pin configuration effects on early secondary displacement in the surgical treatment of pediatric supracondylar humeral fractures (SCHF).

DETAILED DESCRIPTION:
The study consisted of 100 (68M, 32F) children who underwent surgery between 2010 and 2013 for Gartland Type 3 (SCHF). The patients divided into five groups according to the top in configurations (crossed 1 lateral 1 medial, crossed 2 lateral 1 medial, crossed 1 lateral 2 medial, 2 lateral divergent, and 3 lateral divergent). The average age at the time of injury was 7.34 (between 2 and 14 years). Bauman angle (BA), Humerocapital angle (HCA), Anterior humeral line (AHL), flexion range, extension range, and Carrying angle (CA) were compared at preoperative, postoperative 1st-day, postoperative last control, and non-operated side. The mean follow-up time 24,96±11,06 with a range of 12-54 months.

ELIGIBILITY:
Inclusion Criteria

* Pediatric Gartland Type 3 supracondylar humeral fracture
* Patients operated between 2010-2013
* Patients under 16 years old

Exclusion Criteria:

* Pathological fractures
* Conservative treated supracondylar fractures
* Less than the 1-year follow-up
* Patients with incomplete postoperative follow-up
* Patients older than 16 years
* Pediatric Gartland Type 1 and 2 supracondylar humeral fracture

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients under 16 years.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2015-02-20 (Actual)

PRIMARY OUTCOMES:
Baumann Angle | postoperative 1. day, 1. month and 12. month
  This angle is formed by the humeral axis and a straight line through the epiphyseal plate of the capitellum. Preoperative and postoperative angle differences are measured in anteroposterior and lateral X rays. These differences are measured for reduction quality and these parameters shows the success of the surgery.
Anterior Humeral Line | postoperative 1. day, 1. month and 12. month
  A line drawn down the anterior surface of the humerus should intersect the middle third of the capitellum. Preoperative and postoperative angle differences are measured in anteroposterior and lateral X rays. These differences are measured for reduction quality and these parameters shows the success of the surgery.
Humero-Capital Angle | postoperative 1. day, 1. month and 12. month
  On lateral X-ray angle between capitellum and humeral shaft. Preoperative and postoperative angle differences are measured in anteroposterior and lateral X rays. These differences are measured for reduction quality and these parameters shows the success of the surgery.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT04780308/Prot_SAP_000.pdf